CLINICAL TRIAL: NCT06319963
Title: An Open-Label Phase 1/2a Clinical Trial to Evaluate the Safety, Immunogenicity, and Preliminary Efficacy of a Lentiviral Vector-Based Therapeutic Vaccine Against Human Papilloma Virus (Lenti-HPV-07) in Participants With HPV-Associated Oropharyngeal Squamous Cell Cancer or Cervical Cancer
Brief Title: A Study to Evaluate Lenti-HPV-07 Immunotherapy Against HPV+ Cervical or Oropharyngeal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Theravectys S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Lenti-HPV-07-CT01
Record Dates: First submitted 2024-02-27; First posted 2024-03-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: HPV-Related Cervical Carcinoma; HPV Positive Oropharyngeal Squamous Cell Carcinoma
Keywords: HPV16; Cervical Cancer; Oropharyngeal cancer; Immuno-oncotherapy; Head and Neck Cancers; T-cell vaccine; Lentiviral Vector; Anti-tumor immunity; Early E- and E7 antigens; HPV18; Human Papillomavirus
MeSH Terms: conditions — Uterine Cervical Neoplasms; Oropharyngeal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1/2a, open label, multicenter, dose-escalation and dose expansion trial to assess the safety, tolerability, and preliminary efficacy of Lenti-HPV-07 to participants with HPV associated oropharyngeal squamous cell cancer or cervical cancer. Three dose strengths will be investigated: a low, midlevel, and high dose. Lenti HPV-07 will be administered as either 2 × intramuscular (IM) injections to participants in arm A (recurrent or metastatic stage, refractory to previous treatments) or as a single IM injection to participants in Arm B (newly diagnosed with locally advanced HPV+ cancer never treated). Eligible participants in Arm B will receive only 1 injection of Lenti-HPV-07 prior to the initiation of their standard of care (SoC) therapy. After 18 participants in either arm have been treated in the escalation phase and have completed the 14 day DLT period, the Safety Review Committee and Sponsor will determine the OBD for use in the dose expansion phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A : Refractory newly diagnosed (Experimental): Refractory recurrent and/or metastatic cervical or oropharyngeal cancer that is not amenable to local therapy with curative intent (ie, surgery or radiation therapy with or without chemotherapy).
  Interventions: Drug: Two IM injections Lenti-HPV-07
- Arm B : newly diagnosed locally advanced (Experimental): Participants who have newly diagnosed locally advanced HPV-related oropharyngeal cancer (defined by AJCC 8th edition [ie, T1-2N2-N3, T3-T4N0-N3]) or cervical cancer (stages IB to IVA) that has never been treated with curative intent, and who are candidates to begin an SoC treatment (surgery, radiation therapy with or without chemotherapy).
  Interventions: Drug: One IM injection Lenti-HPV-07

INTERVENTIONS:
Drug: Two IM injections Lenti-HPV-07 — two Lenti-HPV-07 intramuscular injections one month apart
  Arms: Arm A : Refractory newly diagnosed
Drug: One IM injection Lenti-HPV-07 — a single intramuscular injection prior to receiving a standard of care 28 days at least after the injection.
  Arms: Arm B : newly diagnosed locally advanced

SUMMARY:
The goal of this clinical trial is to learn about the safety and efficacy of a potential new treatment called Lenti-HPV-07 in patients with a cancer induced by Human Papilloma Virus (HPV).

The main questions aim to answer are:

* Is Lenti-HPV-07 safe?
* Does Lenti-HPV-07 induce an immune response?

Participants will be assigned to a group based on their cancer type

* either study drug group A: recurrent and/or metastatic cancer
* or study drug group B: newly diagnosed with locally advanced cancer

After they finish the study treatment, they will be followed for up to 1 year. Follow-up visits will occur via clinic visits or phone calls 4 weeks after the last study treatment and then quarterly for up to 1 year.

DETAILED DESCRIPTION:
As of 06Nov2025 the recruitment in ARm A of the study (recurrent/metastatic cancers) has been closed to further enrollment, in accordance with the protocol and the study's prespecified operational and/or scientific considerations. No new participants will be enrolled into Arm A, and no additional study drug will be administered within this arm.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed invasive HPV-related oropharyngeal or cervical cancer
* ECOG performance status of 0 or 1
* adequate hepatic, renal, pulmonary, and bone marrow/hematological function

Exclusion Criteria:

- with seropositivity for HIV, active hepatitis C virus (HCV) infection, or hepatitis B (HBV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 12 months after last injection
  Frequency, intensity, and relationship of adverse events with vaccine administration per CTCAE v5.0
OBD | 28 days after last injection
  To identify the optimal biological dose (OBD) and schedule for subsequent trials of Lenti-HPV-07

SECONDARY OUTCOMES:
Immunogenicity | 12 months after last injection
  * measure of CD4+ and CD8+ T cell responses specific to E6 or E7 from HPV16 and HPV18 in PBMC
  * repertoire and clonotype tracking, and cytometric analysis of T cell activation/effector/memory marker
PD-L1 expression | 12 months after last injection
  PD-L1 tumor expression, as measured by composite positive score, by 50% both pre- and post-injection

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Florida Cancer Specialists (from Sarah Canon research Institute), Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: Undecided